CLINICAL TRIAL: NCT03189004
Title: Assessing the Impact of Mobile Phone Technology to Improve Health Nutrition and Population (HNP) Service Utilization in Rural Bangladesh Through Pilot Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PR-16019
Record Dates: First submitted 2017-05-21; First posted 2017-06-16 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Maternal Health; Child Health; Vaccination; Family Planning Services
Keywords: mHealth, health services, technology, smartphones, Bangladesh
MeSH Terms: interventions — Population

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Identification and registration of pregnant women and servic (Active Comparator): Pregnant women will receive auto reminder through their mobile for ANC visit prior to their scheduled date for each visit via voice message followed by text message. The schedule visit date will be calculated by the system automatically from the LMP. The reminder will include the date, time, available facilities and services for ANC, and will be sent to the women several times to ensure their ANC visits. The system will also send auto reminder through text message to the concerned service provider to check whether the pregnant woman has received ANC or not. The service provider will provide and update the ANC services and status of the particular pregnant woman. Apart from ANC reminders, the pregnant women will also receive voice message on healthcare during pregnancy, danger signs and birth preparedness.From the LMP, the expected date of delivery (EDD) will be calculated by the system and reminder will be sent to the pregnant women automatically.
  Interventions: Behavioral: Impact of Mobile Phone Technology to Improve Health Nutrition and Population (HNP) Service Utilization in Rural Bangladesh
- Birth notification (Active Comparator): The pregnant women will be encouraged and trained to notify immediately after the delivery through SMS by themselves or by anyone on behalf of the delivered women. After receiving birth notification, system will automatically update the particulars of newborns including date of birth, PNC schedule, EPI vaccination due dates for the newborn and location of service centre. The system will also send auto reminder to the mothers with a specific time schedule for PNC visit, newborn care visit and schedule of receiving vaccines for the newborn.
  Interventions: Behavioral: Impact of Mobile Phone Technology to Improve Health Nutrition and Population (HNP) Service Utilization in Rural Bangladesh
- Childhood vaccination services under EPI (Active Comparator): After the outcome of the delivery of the registered pregnant women, the system will receive the birth notification as mentioned in the birth notification process. Mothers/caregivers of the newborn will receive auto voice/text messages one day prior to their visit to the vaccination centres. A second reminder will be sent to the parents of all the targeted children through their own phones or their family's numbers collected earlier on the vaccination day at the beginning of the vaccination session for bringing their children for vaccination. A third reminder will be sent to the mothers/caregivers of the children who were not vaccinated after receiving the second reminder as scheduled on that day. The system will also provide auto reminder to the concerned service provider including EPI session wise list of targeted children. The service providers will update the status of vaccination of session using their Smartphone
  Interventions: Behavioral: Impact of Mobile Phone Technology to Improve Health Nutrition and Population (HNP) Service Utilization in Rural Bangladesh
- Newly married couple identification (Active Comparator): The Smartphones will contain specific software for newly married couple registration where some necessary information (names of newly married couple, age, address, LMP, current contraceptive use, future fertility plan and mobile phone number) can be updated and sent to the server. A unique ID number will be automatically created. This unique ID will ensure her to get necessary family planning services within the study area. Based on the information gathered through couple registration process, the system will automatically generate the most suitable family planning options for a couple and send the information to the concerned service providers. The service provider will motivate the client for the most suitable FP method option generated by the system and after taking the consent they provide the method accordingly.
  Interventions: Behavioral: Impact of Mobile Phone Technology to Improve Health Nutrition and Population (HNP) Service Utilization in Rural Bangladesh
- e-Referral (Active Comparator): There will be online referral system for the registered women and their children for ANC, PNC, delivery care, neonatal management, IMCI and other complication management in which healthcare providers from lower facilities can refer a patient to the higher facilities. The women will be identified in the higher facilities by their unique ID. The service providers will enter referral data to the system during the referral process and the patients and providers from higher facilities will get system generated reminders about the referral. The service providers in higher facilities will be able to check the health status and cause of referral using patient's unique ID number from the system and will manage accordingly as well as update the given management to the system. If the referred woman does not visit the referral facility, she will receive repeated reminders auto-generated by the system to comply the referral
  Interventions: Behavioral: Impact of Mobile Phone Technology to Improve Health Nutrition and Population (HNP) Service Utilization in Rural Bangladesh
- e-monitoring (Active Comparator): There will be web based monitoring system to oversee the progress and status of all the activities under this study for policy makers, programme peoples and other supervisors from national to the union levels. All these data will be available in the central database which will be visualized and accessible at all concerned levels through internet in particular website. They can constantly follow up the progression and healthcare delivery system of the respective area and provide regular feedback, when necessary. There will be provision of auto-generation of reports for each and every activity through the system by area and service provider specific.
  Interventions: Behavioral: Impact of Mobile Phone Technology to Improve Health Nutrition and Population (HNP) Service Utilization in Rural Bangladesh

INTERVENTIONS:
Behavioral: Impact of Mobile Phone Technology to Improve Health Nutrition and Population (HNP) Service Utilization in Rural Bangladesh — 1. Identification and registration of pregnant women and services for them
  2. Birth notification
  3. Childhood vaccination services under EPI
  4. Newly married couple identification
  5. e-Referral.
  6. e-monitoring
  Other Names: Assessing the Impact of Mobile Phone Technology to Improve Health Nutrition and Population (HNP) Service Utilization in Rural Bangladesh through Pilot Intervention

SUMMARY:
1. Burden:

   In global perspective, it is estimated that the lives of 150,000 women could be saved each year worldwide with access to sufficient family planning services. It is indicated that only 26 percent women received four or more antenatal care (ANC) visits during their pregnancies, while 67.7 percent received at least one ANC during their pregnancies which are the great challenges for ensuring safe motherhood in the country. As a part of safe motherhood, it is estimated that only 28.8 percent deliveries are being conducted in health facilities in the country. In case of postnatal care (PNC), from 2008 to 2010, only 27 percent of women received PNC for their last deliveries from a medically-trained provider within two days of their delivery. Despite the tremendous success of expanded programme on immunization (EPI) in Bangladesh, a substantial number of children are not fully vaccinated under EPI as data shows 82 percent were fully vaccinated by the age of 12 months.
2. Knowledge gap:

   Use of technology for covering all or major components of primary health care (PHC) is yet to be developed and tested in Bangladesh. Further, no such initiative has yet been taken focusing community clinic (CC) to ensure equity of services in Bangladesh.
3. Relevance:

At present in Bangladesh, the CCs cater the services on family planning, maternal neonatal and child health (MNCH), health education for the rural people by using e-health strategy as the community health care provider (CHCP), newly recruited staff of community clinic are equipped with internet connected laptop service. So, updated technology for updating information, follow up and referral in primary health care can be used to increase the utilization of health services.

Hypothesis (if any):

Use of smart phones by community level healthcare providers will increase utilization of reproductive health (RH) and family planning (FP), MNCH, integrated management of childhood illness (IMCI), EPI and other PHC services at rural communities in Bangladesh.

Objectives:

To develop and test a mechanism as well as assess the impact of mHealth strategy to improve RH and FP, MNCH, IMCI, EPI and other PHC services in rural communities of Bangladesh.

Methods:

The service delivery personnel who are providing the services to the community people at different levels (community clinic, union health and family welfare centre, upazila health complex) will be equipped with smart phones having the facilities for text messages, voice messages as well as internet and data capturing. Training on handling of the smart phones, data capturing and monitoring will be provided to service providers in each upazila. They will be trained to input, edit, verify and monitor the data on different services through the software installed in their smart phones. The community clinic management and support groups will be oriented and motivated on mobile phone based registration, notification and referral to the health facilities.

Outcome measures/variables:

This will be a quasi-experimental pre-post design study and evaluation will be done through comparing antenatal care (ANC), postnatal care (PNC), and contraceptive prevalence rate (CPR) and EPI coverage before and after its implementation in the study versus comparison areas. The study will be conducted over a period of 30 months.

DETAILED DESCRIPTION:
Introduction In Bangladesh, about 2 million new faces are added to the population annually with a growth rate of 1.4% . Last Health Population and Nutrition Sector Development Programme (HPNSDP) of the Ministry of Health and Family Welfare (MOHFW) had set a target of total fertility rate (TFR) of 2.0 and contraceptive prevalence rate (CPR) of 72 by 2016 which is currently 2.3 and 61.2 respectively. It is necessary to increase the age at first birth as data indicates almost half of women giving birth by age 18 and nearly 70% giving birth by age 20. It is indicated that only 26% women received four or more antenatal care (ANC) visits during their pregnancies, while 68% received at least one ANC during their pregnancies which are the great challenges for ensuring safe motherhood in the country. As a part of safe motherhood, it is estimated that only 29% deliveries are being conducted in health facilities in the country. In case of postnatal care (PNC), from 2008 to 2010, only 27 percent of women received PNC for their last birth from a medically-trained provider within two days of their delivery . Despite the tremendous success of EPI in Bangladesh, a substantial number of children are not fully vaccinated under EPI as data shows 82% were fully vaccinated by the age of 12 months. In case of diarrhoea among under 5 years of age, 25% received treatment from a health facility or healthcare providers. Thirty-five percent of the children under 5 years who had acute respiratory infection (ARI) received treatment from a health facility or healthcare providers. More than six of every ten children with fever sought treatment from the private medical sector. Although 90% of children are breastfeed until age 2, as recommended, but 36 percent of children less than age 6 months are out of exclusively breastfed. Though the health indictors in Bangladesh are improving, these rates are behind from the target.

In recent years, mobile phone use in healthcare (mHealth) has emerged to augmented of healthcare services where the population is underserved especially in rural areas . In a systematic review, Tamrat and colleagues (2011) highlighted the scope of mHealth along the stages of the 'continuum of care' for maternal, newborn and child healthcare [8]. mHealth programs are being used for pregnancy tracking, appointment reminders for antenatal care, and SMS-based health education during pregnancy. During the birth, mHealth can be used for point-of-care remote consultation, facilitate referral to health facility; facilitate access to health facility and to promote timely contact with community health workers. For postpartum and newborn care, mHealth can be used for maternal and infant growth monitoring, timely reminders for immunization .

In Bangladesh, mHealth and eHealth initiatives are being implemented by MOHFW and different organizations and donors are supporting to the initiatives. This initiative will complement with existing health systems and contribute to increase effectiveness of HPN services by using mobile phone based technologies.

The Government of Bangladesh has placed a high priority on eHealth, which is reflected in the ICT Policy 2009. The strategic areas/issues relevant to health in the ICT Policy 2009 include the following (Clauses 7.1-7.4 of ICT Policy): 'Improve healthcare delivery management through use of telemedicine and modern technology; create awareness at all levels, including hard-to-reach areas with particular importance in making maternal, child and reproductive care available; ensure quality of care and increase the capacity of health care delivery system'. But use of technology for covering all or major components of primary health care (PHC) is yet to be developed and tested in Bangladesh. Further, no such initiative has yet been taken focusing community clinic (CC) to ensure universal health coverage in Bangladesh.

At present, in Bangladesh, the CCs can cater the services on family planning (FP), maternal neonatal and child health (MNCH) and health education for the rural people by using eHealth strategy as the community health care provider (CHCP) and other staff of CCs are equipped with internet connected laptop service . One recent study findings show that 33% rural married women and 69% of their family members have mobile phones. Therefore, the MOHFW, icddr,b and Ethics Advance Technology Limited (EATL) have taken this initiative to utilize mobile phone technology to improve HPN service in rural areas of Bangladesh. This study will be implemented with the aim to develop and test a mechanism of mHealth strategies as well as assessing the impact in improving reproductive health and family planning, maternal neonatal and child health, integrated management of childhood illness, expanded programme on immunization, and other primary health care services in community level in rural areas of Bangladesh. This is an evidence based research for HPN services using mobile technology and proposed extension of the project and integrated with health system of the Government in Bangladesh.

This study aims to: 1) Improve coverage of ANC, delivery care and PNC; 2) Improve use of family planning services among newly married couples to increase the age at first birth; 3) Improve utilization of MNCH services including EPI services to reduce neonatal mortality rate; 4) Assess acceptability of providing health education regarding family planning, nutrition, breastfeeding; 5) Establish technology based referral linkage of CCs with the higher facilities.

Methods Study design

The study will follow a quasi-experimental pre-post design. Evaluation will be carried-out through comparing ANC, delivery care, PNC, contraceptive prevalence rate (CPR) and EPI coverage before and after its implementation between the study and the comparison areas.

Study area

The study will be conducted in two selected administrative divisions of Bangladesh: one high performing (Rajshahi) division and one low performing (Chittagong) division. Based on the performance of health and family planning indicators, the selected districts are: Natore from the high performing (Rajshahi) division and Cox's Bazar from the low performing (Chittagong) division. In high performing division, one upazila (Bagatipara) of Natore district will be the intervention upazila while Baraigram of the same district will be the comparison upazila. On the other hand, one upazila (Chakaria) of Cox's Bazar district will be the intervention upazila while Ramu will be the comparison upazila. A total of 4 upazilas (2 intervention and 2 comparision upazilas) from the two divisions will be selected for the study.

Timeline The study will be conducted over a period of 30 months in three phases: (i) inception phase (6 months for IRB approval, recruitment of staff, stakeholders' meetings at different levels, mobile apps and survey instrument development, training of GoB staff on interventions, baseline survey and inception report preparation); (ii) intervention implementation phase (18 months for implementation of intervention; (iii) evaluation phase (4 months for end line data collection, data analysis and report writing, sharing of the results and evidence for future scaling up through dissemination, finalization of report and publications).

Mobile apps development and testing

The mobile apps were developed by a team a team from Ethics Advanced Technology Limited (EATL). After developing the apps study team did the filed test and piloting in other than project areas. After receiving the feedback, study team tried to make the easiest apps. The SMS messages were developed by a team comprising of general physicians, immunization expert, family planning expert, health systems expert, health care provider, GoB officials and non government officials. After developing the SMS messages in Bengali, study team sent these messages to several individuals in the pre-test stage including persons who can only read SMS and have no formal education qualifications. After receiving the feedback, study team tried to make the contents of the SMS suitable for the general population. Investigators will ensure that all our participants in the study can read the SMS messages by themselves or someone in the family who can describe the messages to them if they do not understand.

Interventions

The Bangladesh government provides primary health care services to all citizens through a three-tiered healthcare service delivery system: the community clinics, each for 8000 people; the union health and family welfare centres (UH&FWCs), each for 25,000 people; and the upazila (sub-district) health complexes (UHCs) with an out-patient and an emergency departments, 50 in-patient beds and an operating room, each for 250,000 people, which coordinate services between different tiers. The service delivery personnel at different levels (CC, UH&FWC, UHC) will be equipped with Smartphones having the facilities for text messages, voice messages as well as internet and data capturing. Smartphones will be provided to them from the project. Training on handling of the Smartphones, data capturing and monitoring will be provided to upazila Health and family planning officer (UHFPO), upazila family planning officer (UFPO), medical officers (health and family planning departments), the statistical assistant, family welfare visitors (FWVs), sub-assistant community medical officers (SACMOs), nurses and medical technologist, health inspectors (HIs), family planning inspectors (FPIs), assistant health inspectors (AHIs), health assistants (HAs), family welfare assistances (FWAs), community health care providers (CHCPs) and other related service providers in each upazila. They will be trained to input, edit, verify and monitor the data on different services through the software installed in their Smartphones. The community clinic management and support groups will be oriented and motivated on mobile phone based registration, notification and referral to the health facilities. A team from Ethics Advanced Technology Limited (EATL), a software development company will provide technical support to develop the device, train concerned personnel, and continue support in smooth functioning of the system. The interventions to be tested are as below:

1. Identification and registration of pregnant women and services for them

   For fixing the target population for ANC, PNC and delivery care, pregnancy identification and registration is the initial activity. A routinely updated list of all the pregnant women of every village is supposed to be available with all FWAs. However, this list can be updated from information of other service providers like HAs, FWVs, and CHCPs. Pregnant women will be identified and registered in the following ways: from routine community visits of health and family planning workers; from EPI centres when the pregnant mothers visit for receiving TT vaccine; from registers of pregnant mothers with community clinics; from satellite sessions conducted by FWVs; from registers of pregnant mothers maintained by FWVs at UH&FWCs and UHC; from combined meetings held at community clinics, UH&FWC and UHC, and; from registers of pregnant mothers maintained by NGOs who are working on reproductive, maternal and child health.

   Registration process of pregnant women: The Smartphones carried by the healthcare service providers will contain a customize software for registration of pregnant women with information (name of pregnant women, age, address, last menstruation period (LMP) and mobile phone number) and updating and sending to the server. A unique identification (ID) number will be automatically created followed by data upload to the server and will be given to the pregnant women. This unique ID will ensure her to get necessary healthcare services within the study area.

   Service delivery system for ANC, delivery care, essential newborn care and PNC: Pregnant women will receive auto reminder through their mobile for ANC visit prior to their scheduled date for each visit via voice message followed by text message. The schedule visit date will be calculated by the system automatically from the LMP. The reminder will include the date, time, available facilities and services for ANC, and will be sent to the women several times to ensure their ANC visits. The system will also send auto reminder through text message to the concerned service provider to check whether the pregnant woman has received ANC or not. The service provider will provide and update the ANC services and status of the particular pregnant woman. Apart from ANC reminders, the pregnant women will also receive voice message on healthcare during pregnancy, danger signs and birth preparedness.From the LMP, the expected date of delivery (EDD) will be calculated by the system and reminder will be sent to the pregnant women automatically. The pregnant woman will receive auto voice messages/text messages containing necessary information related to institutional delivery according to her EDD.
2. Birth notification

   The pregnant women will be encouraged and trained to notify immediately after the delivery through SMS by themselves or by anyone on behalf of the delivered women. After receiving birth notification, system will automatically update the particulars of newborns including date of birth, PNC schedule, EPI vaccination due dates for the newborn and location of service centre. The system will also send auto reminder to the mothers with a specific time schedule for PNC visit, newborn care visit and schedule of receiving vaccines for the newborn.
3. Childhood vaccination services under EPI

   After the outcome of the delivery of the registered pregnant women, the system will receive the birth notification as mentioned in the birth notification process. Mothers/caregivers of the newborn will receive auto voice/text messages one day prior to their visit to the vaccination centres. A second reminder will be sent to the parents of all the targeted children through their own phones or their family's numbers collected earlier on the vaccination day at the beginning of the vaccination session for bringing their children for vaccination. A third reminder will be sent to the mothers/caregivers of the children who were not vaccinated after receiving the second reminder as scheduled on that day. The system will also provide auto reminder to the concerned service provider including EPI session wise list of targeted children. The service providers will update the status of vaccination of session using their Smartphone and the system will allow the service providers to see the drop-out and left out cases.
4. Newly married couple identification

   Newly married couple identification and registration is the initial activity for fixing the target population for FP service. A routinely updated list of all the newly married couple of every village is supposed to be available with all FWAs. However, this data can be updated from other service providers also, such as HAs, FWVs, CHCPs. Couple identification and registration will be done through following ways: during their regular community visits; from service delivery points like community clinics, UH&FWCs and UHC; at satellite sessions by FWVs; and from other NGOs who are working on reproductive health.

   Newly married couple registration process: The Smartphones will contain specific software for newly married couple registration where some necessary information (names of newly married couple, age, address, LMP, current contraceptive use, future fertility plan and mobile phone number) can be updated and sent to the server. A unique ID number will be automatically created followed by data upload to the server and will be given to the couple. This unique ID will ensure her to get necessary family planning services within the study area.

   Family planning service delivery system:Based on the information gathered through couple registration process, the system will automatically generate the most suitable family planning options for a couple and send the information to the concerned service providers. The service provider will motivate the client for the most suitable FP method option generated by the system and after taking the consent they provide the method accordingly. The system will send auto messages to the couples through their mobile phones about importance of birth spacing and use of FP methods, information related to services at CCs and UH&FWCs. The service provider will update information to the system to maintain the information of FP method use and regular follow up status which will be recorded in server.
5. e-Referral

   There will be online referral system for the registered women and their children for ANC, PNC, delivery care, neonatal management, IMCI and other complication management in which healthcare providers from lower facilities can refer a patient to the higher facilities. The women will be identified in the higher facilities by their unique ID. The service providers will enter referral data to the system during the referral process and the patients and providers from higher facilities will get system generated reminders about the referral. The service providers in higher facilities will be able to check the health status and cause of referral using patient's unique ID number from the system and will manage accordingly as well as update the given management to the system. If the referred woman does not visit the referral facility, she will receive repeated reminders auto-generated by the system to comply the referral; and the service provider who referred the mother/client will be able to see the status of the client using smart phone.
6. e-monitoring

There will be web based monitoring system to oversee the progress and status of all the activities under this study for policy makers, programme peoples and other supervisors from national to the union levels. All these data will be available in the central database which will be visualized and accessible at all concerned levels through internet in particular website. They can constantly follow up the progression and healthcare delivery system of the respective area and provide regular feedback, when necessary. There will be provision of auto-generation of reports for each and every activity through the system by area and service provider specific. Figure-2 shows the interventions implementation process and Figure-3 shows the snap shots of apps developed.

Study population The study populations will be: (i) currently married women of reproductive age not currently pregnant and did not have delivery within last 6 months; (ii). Mothers of children aged 12-23 months for assessing children's vaccination coverage; (iii). Mothers of children aged 0-11 months for assessing ANC, delivery care, PNC and vaccination coverage; and iv. The healthcare service providers.

Procedures for selection of sample clusters: In the catchment area of a CC there are 8 routine EPI centers (including the CCs one) each serving, on an average, ~1000 people (or ~235 households). The catchment area of the EPI centre will be treated as 'cluster'. Given the crude birth rate of ~20 per 1000 population per year there will be 20 mothers who have a infant aged 0-11 months eligible to provide information on ANC, delivery care and PNC; and another 20 mothers who have a toddler aged 12-23 months eligible to provide information on child vaccination. As such, 33 EPI centers from the list of EPI centers of an upazila (with at least one EPI centre per CC) in the selected sub-district will be randomly chosen for survey.

Selection of households: The second stage will be selection of households with eligible respondents in each sampled cluster (or EPI centre catchment area). With their consent all mothers with child aged 0-11 months or 12-23 months will be interviewed for maternity care and vaccination respectively. Women (married non-pregnant or did not delivered baby in <6 months) eligible for family planning use are many in a cluster. Therefore, a woman eligible for family planning method use living in the household next to the mother with a child aged 0-11 months will be interviewed. The same sample selection procedures will be followed in the comparision areas.

ELIGIBILITY:
Inclusion Criteria:

* Currently married women of reproductive age not currently pregnant and did not have delivery within last 6 months
* Mothers of children aged 12-23 months for assessing children's vaccination coverage, and
* Mothers of children aged 0-11 months for assessing ANC, delivery care, PNC and vaccination coverage
* The service providers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5280 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
ANC | Assess the recommend number of ANC (4 ANC) coverage 18 months after intervention
  Number of ANC coverage before and after its implementation
PNC | Assess the recommend number of PNC (3 ANC) coverage 18 months after intervention
  Number of PNC coverage before and after its implementation
Contraceptive prevalence rate (CPR) | Assess the Contraceptive prevalence rate (CPR) at the end of intervention of 18 months.
  Assess the Contraceptive prevalence rate (CPR) coverage
EPI coverage | Assess the EPI vaccination coverage at the end of the intervention of 18 months
  EPI coverage before and after its implementation

CONTACTS AND LOCATIONS:
Overall Officials: Jasim Uddin, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276